CLINICAL TRIAL: NCT05948488
Title: Psychological Study of the Links Between Feeling and Fear of Pain, Anxiety and Quality of Life in Children With Mucoviscidosis
Brief Title: Psychological Study in Children With Mucoviscidosis
Acronym: DoulAnxMuco
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/18/0304; 2018-A02216-49 (Other: ID-RCB)
Record Dates: First submitted 2023-07-05; First posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Children; Pain; Anxiety
MeSH Terms: conditions — Cystic Fibrosis; Pain; Anxiety Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with cystic fibrosis: Children over 8 and under 18 with cystic fibrosis. Children must be represented by their parent.
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — The questionnaires focus on anxiety, fear and quality of life.

SUMMARY:
Cystic fibrosis is the most common serious genetic disease in Europe. It is a multi-disciplinary disease, causing multiple organ damage. It is a painful disease and a source of anxiety and depression.

The aim of this study is to assess the link between pain experienced during care and anxiety in children aged over 8 with cystic fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Have cystic fibrosis
* Child aged over 8 years and under 18 years
* Presence of at least one parent at the time of inclusion
* To be present for a scheduled hospitalisation at the Resources and Competence Centres for Cystic Fibrosis
* Do not object to the research

Exclusion Criteria:

* Under 8 or over 18 years of age
* Lack of at least one parent at the time of inclusion
* Presence of chronic co-morbidities
* Difficulty reading and understanding French
* Objection to taking part in research

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children over 8 and under 18 with cystic fibrosis. Children must be represented by their parent.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2022-08-28 (Actual); Study Completion 2022-08-28 (Actual)

PRIMARY OUTCOMES:
Links between pain during care and anxiety | 1 day
  Pain during care is assessed using the Visual Analogic Scale (VAS) and anxiety using the State Trait Anxiety Inventory (STAI) scale.
  The Visual Analogic Scale (VAS) is a self-assessment scale. It is a line. At one end is indicated: 0 "no pain", at the other: 100 "unbearable pain".
  The State Trait Anxiety Inventory (STAI) is a self-assessment scale. It consists of 20 items. For item, the child has to choose one of three modalities : almost never, sometimes, often. The higher the score, the more severe the anxiety.

SECONDARY OUTCOMES:
Links between pain-related fears and pain during care | 1 day
  Pain related fears is assessed using the Fear of Pain Questionnaire (FOPQ) and pain during care using the Visual Analogic Scale (VAS).
  The Fear of Pain Questionnaire (FOPQ) is a self-assessment scale. It consists of 24 items. For item, there are five modalities : strongly disagree, disagree, don't know, agree, strongly agree.
  The Visual Analogic Scale (VAS) is a self-assessment scale. It takes the form of a line. At one end is indicated: 0 "no pain", at the other: 100 "unbearable pain".
Links between pain during care and quality of life | 1 day
  Pain during care is assessed using the Visual Analogic Scale (VAS) and quality of life using the Cystic Fibrosis Questionnaire (CFQ).
  The Visual Analogic Scale (VAS) is a self-assessment scale. It is a line. At one end is indicated: 0 "no pain", at the other: 100 "unbearable pain".
  The Cystic Fibrosis Questionnaire (CFQ) composed of four modalities : always, often, sometime, never.
Links between pain during care and the severity of the disease | 1 day
  Pain during care is assessed using the Visual Analogic Scale (VAS) and the severity of the disease by the number of respiratory exacerbations per year.
  The Visual Analogic Scale (VAS) is a self-assessment scale. It is a line. At one end is indicated: 0 "no pain", at the other: 100 "unbearable pain".
Links between the severity of the disease and anxiety | 1 day
  Anxiety is assessed using tthe State Trait Anxiety Inventory (STAI) scale and the severity of the disease by the number of respiratory exacerbations per year.
  The State Trait Anxiety Inventory (STAI) is a self-assessment scale. It consists of 20 items. For item, the child has to choose one of three modalities : almost never, sometimes, often. The higher the score, the more severe the anxiety.
Links between parents' anxiety and the child's anxiety | 1 day
  Parent's anxiety and child's anxiety is assessed using tthe State Trait Anxiety Inventory (STAI) scale.
  The State Trait Anxiety Inventory (STAI) is a self-assessment scale. It consists of 20 items. For item, the child has to choose one of three modalities : almost never, sometimes, often. The higher the score, the more severe the anxiety.
  The scale is suitable for parents and children.

CONTACTS AND LOCATIONS:
Overall Officials: Géraldine LABOURET, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Géraldine LABOURET, Toulouse, France